CLINICAL TRIAL: NCT01048619
Title: Phase 1 Study to Assess Tolerability, PK and PD Activity of ON 01910.Na Administered Orally as Escalating Single and Multiple Doses Twice a Day up to 14 Days of a 21-Day Cycle in Patients With Myelodysplastic Syndrome
Brief Title: Safety and Pharmacokinetic Study of Oral ON 01910.Na in Patients With Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Traws Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-01
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Myelodysplastic Syndrome
Keywords: Myelodysplastic Syndrome; MDS
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — ON 01910

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ON 01910.Na (Experimental): The maximum tolerated dose of oral ON 01910.Na administered in a fasting state (defined as no less than 30 min before next meal) twice a day for 14 days will be determined following an adaptive design at doses between 70 and 700mg.
  Interventions: Drug: ON 01910.Na

INTERVENTIONS:
Drug: ON 01910.Na — In Part I, the bioavailability and tolerability of ON 01910.Na as single, oral, escalating doses in a fasting state (defined as no less than 30 min before next meal) is studied. Three patients get 70mg dose the 1st week. In the absence of drug-related grade 2 toxicity or higher, doses will escalate in each patient weekly (wk) to 140mg (wk 2), 280mg (wk 3), 560mg (wk 4) and 700mg (wk 5). At end of Part I all patients will be eligible for Part II. Part II proceeds if drug is measured in plasma and DLT not observed at 70mg dose in Part I. The maximum tolerated dose of oral ON 01910.Na administered in a fasting state (defined as no less than 30 min before next meal) twice a day for 14 days will be determined following an adaptive design at doses between 70 and 700mg.
  Other Names: rigosertib

SUMMARY:
In other clinical studies, ON 01910.Na has been safely given intravenously to Patients with advanced cancers. However, to treat some Patients, it may be better if ON 01910.Na could be given by mouth. This study will determine if it is safe to give ON 01910.Na by mouth, what is the highest dose can be safely given by mouth, and how much of the drug gets from the stomach into the blood stream when it is given by mouth.

DETAILED DESCRIPTION:
This is a three-part phase 1 study in which nineteen to one hundred two patients with Low, Intermediate-1, Intermediate-2, or High risk MDS will receive oral doses of ON 01910.Na Concentrate as escalating single or multiple doses (70mg to 700 mg bid) up to 14 days of a 21-day cycle.

Part I: Bioavailability and Tolerability of Single Oral Dosing (n=3):

In Part I of this trial the bioavailability and tolerability of oral ON1910.Na administered as single, oral, escalating doses in a fasting state (defined as no less than 30 minutes before next meal) will be determined in three patients with Low, Intermediate-1, Intermediate-2 or High Risk MDS. All three patients will receive during the first week a 70mg single oral dose and blood samples for pharmacokinetic analyses will be taken after dosing. In the absence of drug-related grade 2 toxicity or higher, single dosing will be escalated in each patient weekly to 140mg (week 2), 280mg (week 3), 560mg (week 4) and 700mg (week 5).

At the end of Part I (week 6), all patients will be eligible to be enrolled in Part II.

Part II: Determination of MTD (n=10-84):

Part II will proceed if measurable drug levels have been measured in Part I and in the absence of DLT at the 70 mg single dose level in Part I. The maximum tolerated dose of oral ON1910.Na administered in a fasting state (defined as no less than 30 minutes before next meal) twice a day for 14 consecutive days will be determined in patients in patients with Low, Intermediate-1, Intermediate-2 or High Risk MDS following an adaptive design.

If blood levels were detected only at the 560mg or 700mg dose level in Part I, then the starting dose will be 140 mg. If blood levels were detected at the 280mg dose level or below, then the starting dose will be 70mg. Initially, patients will be enrolled in two-patient cohorts.

* In the absence of drug-related grade 2 or higher toxicity in either one of the two patients treated for an entire 21-day first cycle (treated for a complete 14 day-period and followed up for another 7 days), the next two patients will be receiving a dose escalated by 100% from prior dose (e.g. 140mg from 70mg prior dose; next dose levels will be 280, 560 and 700mg).
* If drug-related grade 2 or higher toxicity is observed in at least one of the two patients treated for a full 21-day cycle, the cohort will be expanded in order to obtain 3 evaluable (treated for an entire 21-day first cycle) patients.
* If no dose limiting toxicity (DLT) is observed in the first three patients treated for an entire 21-day first cycle, then the next three patients will be enrolled at a dose level increased by 50% from prior dose (e.g. 105mg from 70mg prior dose; see Table 1 below).
* If one DLT is observed in the first three patients treated for an entire 21-day first cycle, then the three next patients will be enrolled at the same dose level.
* If no more than one DLT is observed in the six patients treated for an entire 21-day cycle, then the next six patients will be administered a dose level increased by 25% from prior dose (e.g. 88mg for 70mg prior dose; see Table 2 below) and all subsequent dose escalations will not exceed 25%.
* If two or more patients in any cohort experience DLT, then the maximum tolerated dose (MTD) will have been exceeded and no further dose escalation will occur. The MTD will be established as the immediate prior dosing level
* Identical rules will be applied to all cohorts of patients recruited to the study.

DLT must be at least possibly attributable to ON 01910.Na and is defined as:

* Grade 3 non-hematological toxicity other than nausea, vomiting, diarrhea, fever, esophagitis/dysphagia
* Grade 3 nausea and vomiting uncontrolled by antiemetics; grade 3 diarrhea uncontrolled by antidiarrheal agents; grade 3 drug-induced fever uncontrolled by antipyretics
* Grade 3 stomatitis and/or esophagitis/dysphagia lasting > 3 days
* Delay in recovery to baseline blood counts below pre-treatment baseline (>20% difference) of more than 30 days in the absence of a response

If a patient has a DLT (see definition above) beyond the completion of the first 21-day cycle, administration of oral ON 01910.Na, treatment will be discontinued or reduced (at the discretion of the Principal Investigator) to the lower dose level, or by 25% if the patient was treated at the 70mg dose level. Patients should return to within 20% of their baseline, pre-cycle ANC, platelet or hemoglobin levels prior to treatment with a subsequent cycle. Treatment can be delayed for up to 21 days (1 cycle length) until counts return to their pre-treatment baseline. If counts are still not adequate for treatment, the patient will be re-evaluated 2 weeks later. If any non-hematological toxicity of Grade 2 or 3 is present on the day of ON 01910.Na administration, the drug administration will be withheld until resolution to ≤ grade 1 toxicity is present.

ON 01910.Na blood concentrations will be determined 1 hours after first dosing on days 1, 7 and 14 in all patients recruited in Part II.

Treatment will be continued until progression or stopped in the absence of bone marrow response or hematological improvement after 16 weeks.

Part III: Food/Fast and Absolute Bioavailability PK analysis at MTD in confirming cohort (n=15):

Up to fifteen patients with Low, Intermediate-1, Intermediate-2 or High Risk MDS will be enrolled at the MTD dose level and treated until progression. The treatment will be stopped in the absence of bone marrow response or hematological improvement after 16 weeks.

A subset of twelve patients will undergo the following procedures:

On Day 1, patients will be dosed with ON 01910.Na 800 mg/m2 IV for 24 hours and pharmacokinetic analysis will be performed

* After a wash-out period of 3 days, patients will be dosed with ON 01910.Na MTD dosing in a fasting state twice a day for 3 days. Pharmacokinetic analysis will be performed on the first (Day 5) day of drug administration. Following an overnight fast of at least 10 hours, patients will be administered ON 01910.Na with 240 mL (8 fluid ounces) of water. No food should be allowed for at least 4 hours post-dose. Water can be allowed as desired except for one hour before and after drug administration. Patients should receive standardized meals scheduled at the same time during the pharmacokinetic evaluations.
* After a second wash-out period of 3 days, patients will be dosed with ON 01910.Na MTD dosing in a fed state (defined as within 30 minutes after prior meal) twice a day for 3 days. Pharmacokinetic analysis will be performed on the first (Day 11) day of drug administration. Following an overnight fast of at least 10 hours, patients should start the meal 30 minutes prior to administration of ON 01910.Na. Patients should eat this meal in 30 minutes or less and ON 01910.Na should be administered 30 minutes after start of the meal with 240 mL (8 fluid ounces) of water. No food should be allowed for at least 4 hours post-dose. Water can be allowed as desired except for one hour before and after ON 01910.Na administration.

Oral dosing at MTD level will resume in a fasting state on Day 1 of the second 21-day cycle (14 days of bid dosing followed by a 7-day off treatment period) until progression is noted. The treatment will be stopped in the absence of bone marrow response or hematological improvement after 16 weeks.

If a patient has a DLT (see definition above) beyond the completion of the first 21-day cycle, administration of oral ON 01910.Na, treatment will be discontinued or reduced (at the discretion of the Principal Investigator) to the lower dose cohort level, or by 25% if the patient was treated at the 70 mg dose level. Patients should return to within 20% of their baseline, pre-cycle ANC, platelet or hemoglobin levels prior to treatment with a subsequent cycle. Treatment can be delayed for up to 21 days (1 cycle length) until counts return to their pre-treatment baseline. If counts are still not adequate for treatment, the patient will be re-evaluated 2 weeks later. If any non-hematological toxicity of Grade 2 or 3 is present on the day of ON 01910.Na administration, the drug administration will be withheld until resolution to ≤ grade 1 toxicity is present.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Diagnosis of MDS confirmed within 6 weeks prior to study entry according to the World Health Organization (WHO) Criteria (see Attachment 1) or the French-American-British (FAB) Classification (see Attachment 2).
* Low, Intermediate 1 or 2 or High Risk MDS according to the IPSS score (see Attachment 3)
* At least one cytopenia (Absolute Neutrophil Count < 1500/µL or Platelet Count <100,000/µL or Hemoglobin <10 g/dL)
* Failure of, or insufficient response to Azacytidine or Decitabine or Lenalidomide or to Erythrocyte Stimulating Agent
* Failed to respond to, relapsed following, or opted not to participate in bone marrow transplantation
* Off all other treatments for MDS (including filgrastim (G-CSF) and erythropoietin) for at least four weeks (only 2 weeks if PROCRITTM is used). Filgrastim (G-CSF) can be used before, during and after the protocol treatment for patients with documented febrile neutropenia (<500/µl)
* ECOG Performance Status 0, 1 or 2 (see Attachment 4)
* Willing to adhere to the prohibitions and restrictions specified in this protocol
* Patient (or his/her legally authorized representative) must have signed an informed consent document indicating that he/she understands the purpose of and procedures required for the study and is willing to participate in the study

Exclusion Criteria:

* Anemia due to factors other than MDS (including hemolysis or gastrointestinal bleeding)
* Hypoplastic MDS (cellularity <10%)
* Any active malignancy within the past year except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix or breast
* History of HIV-1 seropositivity
* Uncontrolled intercurrent illness including, but not limited to symptomatic congestive heart failure, unstable angina pectoris or cardiac arrhythmia
* Active infection not adequately responding to appropriate therapy.
* Total bilirubin > 1.5 mg/dL not related to hemolysis or Gilbert's disease, AST/ALT > 2 X ULN
* Serum creatinine > 1.5 x ULN
* Ascites requiring active medical management including paracentesis, or hyponatremia (defined as serum sodium value of <130 Meq/L).
* Women patients who are pregnant or lactating; Male patients with female sexual partners who are unwilling to follow the strict contraception requirements described in this protocol (see Section 4.4).; Patients who do not agree to use adequate contraceptive [including prescription oral contraceptives (birth control pills), contraceptive injections, intrauterine device (IUD), double-barrier method (spermicidal jelly or foam with condoms or diaphragm), contraceptive patch, or surgical sterilization] before entry and throughout the study; Female patients with reproductive potential who do not have a negative serum or urine beta-HCG pregnancy test at screening
* Major surgery without full recovery or major surgery within 3 weeks of ON 01910.Na treatment start.
* Uncontrolled hypertension (defined as a systolic pressure ³ 160 mm Hg and/or a diastolic pressure ³ 110 mm Hg)
* New onset seizures (within 3 months prior to the first dose of ON 01910.Na) or poorly controlled seizures
* Any concurrent investigational agent or chemotherapy, radiotherapy or immunotherapy
* Treatment with standard MDS therapies or investigational therapy within 4 weeks of starting ON 01910.Na
* Psychiatric illness/social situations that would limit the patient's ability to tolerate and/or comply with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-12; Primary Completion 2014-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Hematologic and non-hematologic toxicities and the maximum tolerated dose (MTD) of orally administered ON 01910.Na given twice a day up to 14 days at doses escalating from 70 mg to 700 mg | 2 years

SECONDARY OUTCOMES:
Characterize pharmacokinetics in a fasting state of ON 01910.Na following administration by the oral route. | 2 years
Determine any food effect on the pharmacokinetics and the absolute bioavailability of ON 01910.Na administered orally. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Rami Komrokji, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute; Azra Raza, MD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Columbia University Medical Center, New York, New York

REFERENCES:
- [Result] Navada SC, Silverman LR. The safety and efficacy of rigosertib in the treatment of myelodysplastic syndromes. Expert Rev Anticancer Ther. 2016 Aug;16(8):805-10. doi: 10.1080/14737140.2016.1209413. Epub 2016 Jul 15. PMID 27400247
- [Result] Garcia-Manero G, Fenaux P. Comprehensive Analysis of Safety: Rigosertib in 557 Patients with Myelodysplastic Syndromes (MDS) and Acute Myeloid Leukemia (AML). Blood Dec 2016, 128 (22) 2011; ASH 2016.